CLINICAL TRIAL: NCT00016731
Title: Adolescence, Puberty, Hormones, and Emotion Regulation: An fMRI Study
Brief Title: Adolescence, Puberty, and Emotion Regulation
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010152; 01-M-0152
Record Dates: First submitted 2001-05-31; First posted 2001-06-01 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-10-18

CONDITIONS: Mood Disorder; Neurobehavioral Manifestation; Healthy
Keywords: Depression; Anxiety; CAH; Adults; FMPP; Emotion; Cushing's Syndrome; Adolescence; Magnetic Resonance Imaging; fMRI; Healthy Volunteer; HV; MRI
MeSH Terms: conditions — Mood Disorders; Neurobehavioral Manifestations; Depression; Anxiety Disorders; Cushing Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to use brain imaging technology to compare how the brains of adolescents and adults are activated during tasks that involve emotional responses.

Evidence suggests that adolescents and adults experience activation in similar brain regions when they engage in tasks that involve the processing of emotional stimuli. However, the degree of task-associated activation may differ between adolescents and adults. This study will use functional magnetic resonance imaging (fMRI) to compare brain activation patterns in adolescents and adults. This study will also be used to develop emotion-evoking fMRI tasks to determine whether there are puberty and age-linked components of brain development.

DETAILED DESCRIPTION:
The goal of this project is to use functional magnetic resonance imaging (fMRI) to compare the degree to which brain regions of adolescents and adults with and without steroid-related endocrine disorders are engaged by tasks involving processing of emotionally salient stimuli. In healthy subjects, based on developmental continuities in the relevant psychological processes, we anticipate considerable similarity across age groups in the topography of brain regions engaged by relevant tasks. However, we hypothesize that developmental differences in cortico-limbic circuits of adolescents and adults will be reflected in patterns of fMRI activation. Specifically, we hypothesize in both adults and adolescents that attention and memory tasks involving the processing of emotionally salient stimuli will engage the amygdala, cingulate gyrus, and association cortex of medial/inferior prefrontal cortex and temporal regions. Nevertheless, height of task-associated activation is hypothesized to differ between adolescents and adults within these regions. Moreover, prior studies distinguish puberty vs. age-related aspects of cognitive development: some aspects of attention or memory development relate to changes in chronological age whereas other aspects, particularly those involving emotional processes, relate to pubertal status. Therefore, we expect eventually to use emotion-evoking fMRI tasks to test hypotheses on the presence of complementary, distinguishable puberty vs. age-related components of brain development. In patients with endocrine disorders, we expect to identify abnormal brain function related to defects in steroidogenesis, including in utero hyperandrogenism and hypocortisolism seen in Congenital Adrenal Hyperplasia (CAH), congenital male hyperandrogenism seen in familial male precocious puberty (FMPP), and hypercortisolism seen as Cushing's Syndrome (CS).

To meet these initial goals, we developed and tested a number of attention/emotion tasks in healthy adults and healthy adolescents, tested systematically a few of these tasks in the fMRI, including a face-emotion processing task, an affective picture- processing task, a threat bias task, a dot-probe task, a reward-related task, and tasks probing social processing. We are now entering the 2nd phase of the protocol, in which we are focusing on endocrine disorders, CAH, FMPP and CS. We hypothesize that both face-emotion processing task, an affective picture- processing task will engage the amygdala, cingulate gyrus, and association cortices of the medial/inferior prefrontal and temporal regions differently as a function of time of occurrence, severity, and type of endocrine abnormalities.

ELIGIBILITY:
* INCLUSION CRITERIA: HEALTHY SUBJECTS:

Age: 9-25 (adolescents/young adults); 25-35 (adults).

Consent: can give consent/assent. Parents will provide consent for all minors.

IQ: all subjects will have an IQ greater than 70; assessment relies on WASI.

Psychopathology: all subjects will be free of any current psychiatric disorder as well as lifetime history of psychosis, pervasive developmental disorder, major affective disorder, panic disorder, obsessive compulsive disorder, conduct disorder, ADHD, and anorexia. Assessment relies on comprehensive psychiatric interview.

INCLUSION CRITERIA: ENDOCRINE AND CARRIER PATIENTS

Age: 9-25 (adolescents/young adults); 25-35 (adults).

Consent: can give consent/assent. Parents will provide consent for all minors.

IQ: all subjects will have an IQ greater than 70. Assessment relies on WASI

EXCLUSION CRITERIA:

Any medical condition that increases risk for MRI (e.g. pacemaker, metallic foreign body in eye)

Pregnancy

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2001-05-29; Study Completion 2017-10-18

CONTACTS AND LOCATIONS:
Overall Officials: Monique Ernst, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Weissman MM, Bland RC, Canino GJ, Faravelli C, Greenwald S, Hwu HG, Joyce PR, Karam EG, Lee CK, Lellouch J, Lepine JP, Newman SC, Oakley-Browne MA, Rubio-Stipec M, Wells JE, Wickramaratne PJ, Wittchen HU, Yeh EK. The cross-national epidemiology of panic disorder. Arch Gen Psychiatry. 1997 Apr;54(4):305-9. doi: 10.1001/archpsyc.1997.01830160021003. PMID 9107146
- [Background] Kessler RC, McGonagle KA, Zhao S, Nelson CB, Hughes M, Eshleman S, Wittchen HU, Kendler KS. Lifetime and 12-month prevalence of DSM-III-R psychiatric disorders in the United States. Results from the National Comorbidity Survey. Arch Gen Psychiatry. 1994 Jan;51(1):8-19. doi: 10.1001/archpsyc.1994.03950010008002. PMID 8279933
- [Background] Pine DS, Cohen P, Gurley D, Brook J, Ma Y. The risk for early-adulthood anxiety and depressive disorders in adolescents with anxiety and depressive disorders. Arch Gen Psychiatry. 1998 Jan;55(1):56-64. doi: 10.1001/archpsyc.55.1.56. PMID 9435761